CLINICAL TRIAL: NCT03380871
Title: An Open-Label, Phase 1B Study of NEO-PV-01 With Pembrolizumab Plus Chemotherapy in Patients With Advanced or Metastatic Nonsquamous Non-small Cell Lung Cancer
Brief Title: A Personal Cancer Vaccine (NEO-PV-01) With Pembrolizumab and Chemotherapy for Patients With Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech US Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: BioNTech SE (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-002; KEYNOTE: MK-3475-779
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Cancer; Nonsquamous Nonsmall Cell Neoplasm of Lung
Keywords: Personal Vaccine; Neoantigen; Immunotherapy; Poly-ICLC; Peptide; Checkpoint Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab; Adjuvants, Pharmaceutic; poly ICLC; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NEO-PV-01/Adjuvant + pembrolizumab + chemotherapy (Experimental): Pembrolizumab at a dose of 200 mg administered by intravenous infusion (IV) plus chemotherapy with carboplatin (AUC 5) + pemetrexed (500 mg/m2) every 3 weeks for 4 cycles. At Week 12, all patients, regardless of their disease status, will receive NEO-PV-01 + adjuvant administered subcutaneously (one vial of pooled peptides per injection site) in up to four distinct sites (each extremity or flanks) while continuing therapy with pembrolizumab.
  Interventions: Biological: NEO-PV-01; Biological: Pembrolizumab; Other: Adjuvant; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Biological: NEO-PV-01 — Personal Cancer Vaccine
Biological: Pembrolizumab — monoclonal antibody against PDL1
  Other Names: KEYTRUDA
Other: Adjuvant — immune adjuvant
  Other Names: Hiltonol; Poly-ICLC
Drug: Carboplatin — chemotherapy
Drug: Pemetrexed — chemotherapy
  Other Names: ALIMTA

SUMMARY:
The purpose of this study is to find out if treatment with NEO-PV-01 in combination with pembrolizumab and chemotherapy (pembrolizumab/chemotherapy) is safe and useful for patients with lung cancer. The study also will assess if the NEO-PV-01 vaccine, when given together with pembrolizumab and chemotherapy, can improve your response compared with pembrolizumab and chemotherapy treatment alone. All eligible patients will receive NEO-PV-01 + Adjuvant, pembrolizumab and chemotherapy while on this trial.

DETAILED DESCRIPTION:
This clinical trial will enroll patients with advanced or metastatic nonsquamous non-small cell lung carcinoma not having received treatment for metastatic disease. The five agents being used in this study are:

* A new, investigational, personalized cancer vaccine called "NEO-PV-01"
* Poly-ICLC (Hiltonol), an investigational adjuvant that is used to help stimulate the immune system
* A cancer drug called pembrolizumab (KEYTRUDA®)
* A chemotherapy called pemetrexed (ALIMPTA®)
* A chemotherapy called carboplatin

Both NEO-PV-01 and pembrolizumab are considered immunotherapies and work using the immune system to fight cancer. NEO-PV-01 is a custom made vaccine for you that is based on the specific targets on your cancer. Poly-ICLC is an adjuvant that helps stimulate the immune system and make the vaccine, NEO-PV-01, more effective.

Pembrolizumab helps T-cells, a certain type of immune cell, that recognize these targets to reach and attack your cancer. Pembrolizumab, which is approved in the USA and some other countries, is available by prescription to treat several different cancers, including the type of cancer that you have. Recently, the FDA also approved the combination of Pembrolizumab with chemotherapy for the treatment of your type of lung cancer. This combination works better than each of the drugs on their own.

The purpose of this study is to find out if treatment with NEO-PV-01 in combination with pembrolizumab and chemotherapy is safe and useful for patients with lung cancer. The study also will assess if the NEO-PV-01 vaccine, when given together with pembrolizumab and chemotherapy, can improve your immune response compared with pembrolizumab and chemotherapy treatment alone. The side effects of NEO-PV-01, pembrolizumab, and chemotherapy will be monitored and additional research tests will be done to assess your immune response to your cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Have histologically confirmed unresectable or metastatic nonsquamous NSCLC and having received no prior systemic therapy for metastatic disease.
* Have at least 1 site of disease measurable by RECIST v1.1 that has not been treated with local therapy within 6 months of study treatment. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* At least 1 site of disease must be accessible to provide repeat biopsies for tumor tissue for sequence and immunological analysis. This site may be a target lesion as long as it will not be made unmeasurable by the biopsy procedure.
* Have ECOG PS of 0 or 1 with an anticipated life expectancy of > 6 months.
* Recovered from all toxicities associated with prior treatment to acceptable baseline status (for laboratory toxicities see below limits for inclusion) or a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03, Grade of 0 or 1, except for toxicities not considered a safety risk (eg, alopecia or vitiligo).
* Screening laboratory values must meet the following criteria and should be obtained within 30 days (or 45 days if a biopsy is repeated) prior to study treatment:

  1. White blood cell (WBC) count ≥ 3 × 10e3/µL
  2. Absolute neutrophil count (ANC) ≥ 1.5 × 10e3/µL
  3. Platelet count ≥ 100 × 10e3/µL
  4. Hemoglobin > 9 g/dL
  5. Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 40 mL/min/1.73 m2
  6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for patients with liver metastases
  7. Total bilirubin ≤ 1.5 × ULN (except in patients with Gilbert Syndrome who can have total bilirubin < 3.0 mg/dL). Direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 × ULN.
  8. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  9. Activated Partial Thromboplastin Time (aPTT) ≤1.5 × ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female patients of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 6.4.5.3, for the course of the study through 120 days after the last dose of study medication. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
* Male patients of childbearing potential must agree to use an adequate method of contraception as outlined in Section 6.4.5.3, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of first dose of treatment.
* Received any systemic therapy for cancer treatment including immunotherapeutic agents such as anti-PD1 or anti-PD-L1 antibody therapy.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (ie, ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 30 days prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  1. Note: Subjects with ≤ Grade 2 neuropathy or ≤ Grade 2 alopecia are an exception to this criterion and may qualify for the study.
  2. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients may not receive or have received any radiation therapy at the biopsy sites.
* Received radiation therapy to the lung > 30 Gy within 6 months of first dose of study treatment.
* Received prior tyrosine kinase inhibitor therapy or palliative radiation within 7 days of first dose of study treatment.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging (using the identical imaging modality for each assessment, either MRI or CT scan) for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Patients may not receive any non-oncology vaccine therapy during the period of NEO PV-01 or pembrolizumab administration and until at least 8 weeks after the last dose of the booster vaccine. Seasonal influenza vaccines are allowed but may not be administered between the first dose of pembrolizumab and the last booster dose of NEO-PV-01
* Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF or recombinant erythropoietin) within 4 weeks prior to study Day 1.
* Has active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
* Received a live-virus vaccination within 30 days of planned treatment start.
* Have symptomatic ascites or pleural effusion.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a history of interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Have an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring treatment, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
* Have any underlying medical condition, psychiatric condition, or social situation that, in the opinion of the Investigator, would compromise study administration as per protocol or compromise the assessment of AEs.
* Have a planned major surgery.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* Nursing women are excluded from this study because there is an unknown but potential risk of AEs in nursing infants secondary to treatment of the mother with pembrolizumab, personalized neoantigen peptides, and adjuvant.
* Have a history of an invasive metastatic disease, except for the following:

  1. Individuals with a history of invasive metastatic disease are eligible if they have been disease free for at least 2 years and are deemed by the Investigator to be at low risk for recurrence of that metastatic disease;
  2. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Patients with nonsquamous NSCLC having functionally significant anaplastic lymphoma kinase (ALK) translocations or epidermal growth factor receptor (EGFR) mutations who have not received prior treatment with ALK or EGFR inhibitor.
* Have severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
The rate of adverse events and severe adverse events leading to treatment discontinuation | Baseline through 90 days after the last dose of pembrolizumab
  Rate of adverse events and severe adverse events leading to treatment discontinuation and those adverse events and severe adverse events detected during symptom-directed physical examinations (changes in safety laboratory evaluations, physical examination findings. vital signs, and ECOG PS)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline through 104 weeks
  Objective Response Rate (ORR), defined as the proportion of patients who achieve complete response (CR) or partial response (PR) based on Response Criteria in Solid Tumors (RECIST) v1.1
Clinical Benefit Rate | Baseline through 104 weeks
  Clinical Benefit Rate (CBR), defined as the proportion of patients who achieve a CR, PR, or stable disease (SD) based on RECIST v1.1
Duration of Response | Baseline through 104 weeks
  Duration of Response, DOR, defined as the date of the first documentation of a confirmed response to the date of the first documented PD based on RECIST v1.1
Response Conversion Rate | Baseline to 104 weeks
  Response Conversion Rate (RCR), defined as the proportion of patients who improve in RECIST v1.1 category subsequent to vaccination (eg. PD to SD/PR/CR, SD to PR/CR, PR/CR).
Progression Free Survival | Baseline through 104 weeks
  Progression Free Survival (PFS), defined as the time from the date of first dosing to the date of first documented PD or death
Overall Survival | Baseline of pembrolizumab through 104 weeks
  Overall Survival (OS), defined from the date of enrollment and death from any cause

OTHER OUTCOMES:
T Cell Immune Responses | Day 1 of pembrolizumab/chemotherapy through 104 weeks
  Antigen-specificity in peripheral CD8+ and CD4+ T cell responses following treatment with NEO-PV-01, pembrolizumab, and chemotherapy.
Analysis of Tumor Biopsies | Day 1 of pembrolizumab/chemotherapy through 104 weeks
  Analysis of tumor biopsies following treatment of NEO-PV-01, pembrolizumab, and chemotherapy
Overall Response Rate | Baseline through 104 weeks
  To determine the anti-tumor activity, as assessed by ORR by iRECIST
Progression Free Survival | Baseline through 104 weeks
  To determine the anti-tumor activity, as assessed by PFS by iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Mark DeMario, MD, Study Director — BioNTech US Inc.
Locations (5):
- United States (5):
  - University of California - Los Angeles, Santa Monica, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No